CLINICAL TRIAL: NCT01108432
Title: Hygienists Internet Tobacco Cessation Study (HiQuit)
Brief Title: DPBRN Hygienists Internet Quality Improvement in Tobacco Cessation (HiQuit)
Acronym: HiQuit
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: University of Alabama at Birmingham (Other); University of Massachusetts, Worcester (Other); HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122286; U01DE016747 (NIH)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Smoking Cessation
Keywords: Tobacco cessation counseling
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic Referrals (Experimental): Dental practices randomized to the experimental group will have options on how to refer patients to the tobacco cessation website.
  Interventions: Other: Electronic Referral
- Routine Referral (No Intervention): Dental practices in this arm will refer patients to the Decide2Quit website by using an information prescription.

INTERVENTIONS:
Other: Electronic Referral — Dental practices in this arm will be able to have option of making electronic patient referrals to the Decide2Quit website.
  Arms: Electronic Referrals

SUMMARY:
Our overall goal is to advance science related to using the Internet in health services delivery, and specifically smoking cessation by targeting dental hygienists. Our proposed intervention is the first Internet-delivered intervention to target the dental microsystem for smoking cessation-providing access to hygienists and patients.

DETAILED DESCRIPTION:
This study is designed to allow dental hygienists and dentists to provide additional tobacco cessation counseling with little additional marginal effort. This would be done using an Internet-based referral to external resources. This system, termed "ReferASmoker", will allow hygienists and dentists to refer patients to a patient education, self-management website, "Decide2Quit" and accompanying Quitline, while the patient is still in the dental office. We anticipate that hygienists will be the primary drivers of this intervention. Our intervention has several innovations designed to support the dental practice in their tobacco cessation activities and maximize patient cessation rates. We will randomize 80 community-based primary dental practices into a clinical trial.

Aim 1. To test hypothesis 1(H1)that the number of patients REFERRED to the self-management resource website will be larger in the intervention practices compared to control practices.

Aim 2. To test hypothesis 2 (H2) that the proportion of patients referred who GO to the patient self-management website will be larger in intervention practices compared to control practices

Aim 3. To test hypothesis 3 (H3) that the proportion of smokers who are referred who QUIT at six months will be larger among intervention compared to control because of the additional connectivity of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Community-based practices with internet access available in the office seeing an average of five or more smokers in a week.

Exclusion Criteria:

* Exclude practices that have ongoing computer-based smoking cessation programs for patients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of smokers referred to tobacco cessation website | 12 months
  We will asses the number of patient referrals that the dental hygienists make to the tobacco cessation website.

SECONDARY OUTCOMES:
Proportion of smokers who go to the tobacco cessation website | 12 months
  We will assess the proportion of smokers who were referred to the tobacco cessation website to the number of patients who registered on the website.
Point prevalence smoking cessation | 6 months
  Tobacco cessation behaviors will be assessed by follow-up email and/or telephone interviews at six months from website enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H. GIlbert, DDS, MBA, Study Chair — Dental Practice-Based Research Network (DPBRN); Midge N. Ray, RN, MSN, CCS, Principal Investigator — University of Alabama School of Health Professons at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Health Partners Research Foundation, Minneapolis, Minnesota

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- [Derived] Ray MN, Funkhouser E, Williams JH, Sadasivam RS, Gilbert GH, Coley HL, Rindal DB, Houston TK; National Dental PBRN Collaborative Group. Smoking-cessation e-referrals: a national dental practice-based research network randomized controlled trial. Am J Prev Med. 2014 Feb;46(2):158-65. doi: 10.1016/j.amepre.2013.10.018. PMID 24439349
- [Derived] Coley HL, Sadasivam RS, Williams JH, Volkman JE, Schoenberger YM, Kohler CL, Sobko H, Ray MN, Allison JJ, Ford DE, Gilbert GH, Houston TK; National Dental PBRN and QUITPRIMO Collaborative Group. Crowdsourced peer- versus expert-written smoking-cessation messages. Am J Prev Med. 2013 Nov;45(5):543-50. doi: 10.1016/j.amepre.2013.07.004. PMID 24139766